CLINICAL TRIAL: NCT05712109
Title: Changes in the Force-velocity Relationship of Knee Muscles After ACL Reconstruction
Acronym: FoVeA
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: FoVeA
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2023-03

CONDITIONS: Anterior Cruciate Ligament Injuries; Muscle Weakness
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACL group: The patients were referred to the sport medicine department for the post ACL-R follow-up including isokinetic knee muscle strength evaluations at 4 months and 8 months after the surgery
  Interventions: Other: Follow-up after Anterior cruciate ligament reconstruction

INTERVENTIONS:
Other: Follow-up after Anterior cruciate ligament reconstruction — The patients were referred to the sport medicine department for the post ACL-R follow-up including isokinetic knee muscle strength evaluations at 4 months and 8.months after the surgery

SUMMARY:
Anterior cruciate ligament (ACL) tear is a frequent and devastating injury in sport, especially in pivoting-contact disciplines. In many cases, athletes will undergo an ACL reconstruction (ACL-R) for recovering knee stability, preventing further injuries and returning to sport (RTS). Among the criteria for RTS, knee muscle strength is the most used objective criteria and especially the symmetry of knee flexors and/or extensors between the operated and uninjured knee.

Isokinetic testing of knee muscle strength is considered as a reference for knee muscle testing during the follow up stages after ACL-R. This evaluation allows to measure the strength (torque) of knee flexors and extensors at several angular velocities. However, there is no relevant litterature about the force-velocity (Fo-v) relationship of knee flexors and extensors after ACL-R.

The present study aimed to evaluate and test the differences between the Fo-v relationship parameters between the operated and uninjured knees at 4 months and 8 months after ACL-R, using the 2-points method with isokinetic testing. Also, the investigators aimed to test the impact of the type of surgery (patellar tendon autograft vs. hamstring tendon autograft) on the Fo-v relationship after ACL-R

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had an ACL reconstruction surgery (isolated or associated with other meniscal or ligamentary surgery)
* Patient included in the sport medicine follow-up protocole with intermediate and final isokinetic muscular assessment at 4 months and8 months after surgery respectively
* Patients who completed both tests at the 60°/s and 240°/s velocities

Exclusion Criteria:

* Patient who did not participate in all follow-up consultations and isokinetic muscular assessments
* Cognitive or sensory impairment making it impossible to understand the information form
* Neurological, traumatic or osteoarticular history responsible for muscle imbalance prior to surgery

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All sports patients included in the sport medicine follow-up protocole with isokinetic muscular assessment at 4 months and 8 months after ACL reconstruction surgery since January 2017
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Change in strength | Time Frame: ACL group: Two evaluations on both injured and healthy knees: (1) 4 months after surgery and (2) 8 months after surgery; Routine practice following guidelines
  Measurement of knee extensors and flexors peak strength (in newton.meter, Nm) on isokinetic dynamometer at two angular velocities of 60°/s and 240°/s respectively
Change in the force-velocity relationship | Time Frame: ACL group: Two evaluations on both injured and healthy knees: (1) 4 months after surgery and (2) 8 months after surgery; Routine practice following guidelines
  Calculation of the corresponding slope and maximal force (Y-intercept) of the regression line of the force-velocity curve

SECONDARY OUTCOMES:
Individual characteristics | Time Frame: ACL group: Two evaluations on both injured and healthy knees: (1) 4 months after surgery and (2) 8 months after surgery; Routine practice following guidelines
  Personal characteristics recorded in the medical report as age, gender, type of sport and sport level of practice and return to sport after the surgery
Injury characteristics | Time Frame: ACL group: Two evaluations on both injured and healthy knees: (1) 4 months after surgery and (2) 8 months after surgery; Routine practice following guidelines
  Injury characteristics recorded in the medical report as the type of injury (ACL only, ACL and meniscus, ACL with other ligament injury, recurrent ACL injury) the time before surgery, the type of rehabilitation before and after surgery
Surgery characteristics | Time Frame: ACL group: Two evaluations on both injured and healthy knees: (1) 4 months after surgery and (2) 8 months after surgery; Routine practice following guidelines
  Surgery characteristics recorded in the medical report as the type of surgery, the surgery duration and tourniquet time

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France